CLINICAL TRIAL: NCT03288584
Title: The Effect of Inhibition of Interleukin-6 Activity on Vascular, Endothelial and Left Ventricular Function in Patients With Rheumatoid Arthritis
Brief Title: Effects of Interleukin-6 Inhibition on Vascular, Endothelial and Left Ventricular Function in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Ignatios Ikonomidis, Associate Professor of Cardiology, University of Athens
Other Study IDs: RA-IL6-ATTIKON
Record Dates: First submitted 2017-09-16; First posted 2017-09-20 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Rheumatoid Arthritis; Inflammation
Keywords: Arterial stiffness; Endothelial function; Endothelial glycocalyx; Left ventricular function; Apoptosis; Oxidative stress
MeSH Terms: conditions — Arthritis, Rheumatoid; Inflammation | interventions — tocilizumab; Adrenal Cortex Hormones

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Tocilizumab: Inhibition of Interleukin-6 activity by tocilizumab (Actemra®) 150mg od, sc injection
  Interventions: Drug: Tocilizumab (Actemra®)
- Other biological agent: Other biological agent (TNFa inhibitor, abatacept, rituximab, IL-1Ra)
  Interventions: Drug: Other biological agent
- Corticosteroid and non-biological agents.: Enhanced treatment with corticosteroid and non-biological agents.
  Interventions: Drug: Corticosteroid and non-biological agents.

INTERVENTIONS:
Drug: Tocilizumab (Actemra®) — Inhibition of Interleukin-6 activity by tocilizumab (Actemra®) 150mg od, sc injection
  Groups: Tocilizumab
Drug: Other biological agent — Other biological agent (TNFa inhibitor, abatacept, rituximab, IL-1Ra)
  Groups: Other biological agent
Drug: Corticosteroid and non-biological agents. — Enhanced treatment with corticosteroid and non-biological agents.
  Groups: Corticosteroid and non-biological agents.

SUMMARY:
Recent studies show beneficial effect of the inhibition of interleukin-6 (IL-6) activity on vascular and left ventricular (LV) function. The purpose of this study is to investigate whether anakinra, an IL-6 receptor antagonist, improves vascular, endothelial and LV function in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The inflammatory processes observed in patients with rheumatoid arthritis (RA) are strongly linked to enhanced interleukin-6 (IL-6) activity. Increased IL-6 activity causes myocardial cell damage and endothelial dysfunction. The adverse effects of IL-6 on myocardial and endothelial cells are mediated by an enhanced nitrooxidative stress and the promotion of apoptotic cardiomyocyte death through increased nitrooxidative stress and inflammation. Tocilizumab, a recombinant form of human IL-6 receptor antagonist, is commonly used for the treatment of RA. However it has not been defined whether inhibition of IL-6 activity by tocilizumab shows beneficial effects on endothelial, coronary, arterial and LV systolic and diastolic function in patients with RA.

For this purpose, we studied 60 patients with RA (American Rheumatism Association criteria). All the above subjects had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and corticosteroids and were going to initiate treatment with IL-6 activity inhibitor (tocilizumab). All patients were on treatment with statins and cardioactive medications respectively, for the last 6 months.

All patients were randomized to receive a single injection of tocilizumab (150 mg s.c.), or other biological agent (TNFa inhibitor, abatacept, rituximab, IL-1Ra) or enhanced treatment with corticosteroid and non-biological agents.

Twenty asymptomatic subjects matched for age and sex as the RA patients and with a normal ECG, echocardiogram, and treadmill test were selected as healthy control subjects among subjects attending the cardiology outpatients' clinic.

At baseline in all RA subjects and controls as well as 3 months after the single injection of tocilizumab in RA subjects, we assessed the following parameters a)carotid-femoral pulse wave velocity (PWV), b) the LV dimensions,fractional shortening and wall motion score index (WMSI) c) the systolic (Sm), early diastolic (Em) and late diastolic (Am) myocardial velocities of the mitral annulus by using of tissue Doppler (TDI) as well as the ratio of E wave of the mitral inflow measured by pulsed wave Doppler to the mean Em as an index of LV diastolic filling pressures d) the LV longitudinal, circumferential and radial strain and strain rate, as well as Global Longitudinal strain and Torsion using speckle tracking echocardiography e) the coronary flow reserve (CFR)after adenosine infusion to assess coronary vasomotor function f) the flow-mediated endothelial-dependent dilation of the brachial artery (FMD) to assess peripheral endothelial function g) the diameters of aorta at systole and diastole to calculate the aortic strain as an index of local aortic properties, h) perfused boundary region (PBR) of the sublingual arterial microvessels (ranged from 5-25μm) using Sideview, Darkfield imaging (Microscan, Glycocheck). Increased PBR is considered an accurate index of reduced endothelial glucocalyx thickness because of a deeper red blood cells (RBC) penetration in the glucocalyx. At the same time periods, we measured in blood samples a) nitrotyrosine (NT), protein carbonyls (PC) and malondialdehyde (MDA) to assess oxidative stress, b) soluble Fas and Fas-ligand to assess apoptosis, and c) interleukin-6 and tumor necrosis factor-a to assess inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rheumatoid arthritis who had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and corticosteroids and were going to initiate treatment with interleukin-6 inhibitor.

Exclusion Criteria:

* Familiar hyperlipidemia
* Diabetes mellitus
* Chronic obstructive pulmonary disease or asthma
* Moderate or severe valvular heart disease
* Primary cardiomyopathies
* Malignant tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with rheumatoid arthritis who had an inadequate response to disease modifying antirheumatic drugs (DMARDs) and corticosteroids and were going to initiate treatment with interleukin-6 inhibitor.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-10-27 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Reduction of pulse wave velocity after treatment with tocilizumab | 3 months after treatment
  Reduction of pulse wave velocity (PWV, m/sec) using tonometry after administration of tocilizumab
Increase of global longitudinal strain after treatment with tocilizumab | 3 months after treatment
  Increase of left ventricular global longitudinal strain (GLS, %) using speckle tracking echocardiography after administration of tocilizumab

SECONDARY OUTCOMES:
Reduction of malondialdehyde after treatment with tocilizumab | 3 months after treatment
  Reduction of malondialdehyde (MDA, nmol/L) using spectrophotometry after treatment with tocilizumab
Reduction of protein carbonyls after treatment with tocilizumab | 3 months after treatment
  Reduction of protein carbonyls (PCs, nmol/mg protein) using spectrophotometry after treatment with tocilizumab
Increased of endothelial glycocalyx thickness after treatment with tocilizumab | 3 months after treatment
  Increased of endothelial glycocalyx thickness as assessed by perfused boundary region (PBR, micrometers) of the sublingual arterial microvessels after treatment with tocilizumab

CONTACTS AND LOCATIONS:
Overall Officials: Ignatios Ikonomidis, MD, Principal Investigator — National and Kapodistrain University of Athens
Locations (1):
- Attikon Hospital, Athens, Haidari, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ikonomidis I, Pavlidis G, Katsimbri P, Lambadiari V, Parissis J, Andreadou I, Tsoumani M, Boumpas D, Kouretas D, Iliodromitis E. Tocilizumab improves oxidative stress and endothelial glycocalyx: A mechanism that may explain the effects of biological treatment on COVID-19. Food Chem Toxicol. 2020 Nov;145:111694. doi: 10.1016/j.fct.2020.111694. Epub 2020 Aug 18. PMID 32822775
- [Derived] Ikonomidis I, Pavlidis G, Katsimbri P, Andreadou I, Triantafyllidi H, Tsoumani M, Varoudi M, Vlastos D, Makavos G, Kostelli G, Betaenas D, Lekakis J, Parissis J, Boumpas D, Alexopoulos D, Iliodromitis E. Differential effects of inhibition of interleukin 1 and 6 on myocardial, coronary and vascular function. Clin Res Cardiol. 2019 Oct;108(10):1093-1101. doi: 10.1007/s00392-019-01443-9. Epub 2019 Mar 11. PMID 30859382